CLINICAL TRIAL: NCT04099966
Title: Allogeneic Stem Cell Transplantation for Malignant and Non-malignant Hematologic Diseases Utilizing Alpha/Beta T Cell and CD19+ B Cell Depletion - NYMC 588
Brief Title: AlloSCT for Malignant and Non-malignant Hematologic Diseases Utilizing Alpha/Beta T Cell and CD19+ B Cell Depletion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mitchell Cairo (Other)
Responsible Party: Sponsor-Investigator, Mitchell Cairo, Co-Investgiator, New York Medical College
Organization: New York Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 588
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Leukemia; Severe Aplastic Anemia; Non-hodgkin Lymphoma; Hodgkin Lymphoma; Kostmann; Diamond Blackfan Anemia; Amegakaryocytic Thrombocytopenia; Sickle Cell Disease; Beta-Thalassemia
Keywords: allogeneic stem cell transplantation; t-cell depletion; alpha beta cell depletion
MeSH Terms: conditions — Anemia, Aplastic; Lymphoma, Non-Hodgkin; Hodgkin Disease; Neutropenia, Severe Congenital, Autosomal Recessive 3; Anemia, Diamond-Blackfan; Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- alpha beta cell depletion (Experimental): Matched allogeneic donor stem cells will be processed utilizing α/β CD3+/CD19+ cell depletion with the Prodigy system. Standard pre-conditioning and post-transplant motioning will be given.
  Interventions: Drug: alpha beta depletion

INTERVENTIONS:
Drug: alpha beta depletion — donor cells will be collected and subsequently undergo α/β CD3+/CD19+ cell depletion.
  Other Names: α/β CD3+/CD19+ cell depletion

SUMMARY:
Children, adolescents, and young adults with malignant and non-malignant conditionsundergoing an allogeneic stem cell transplantation (AlloSCT) will have the stem cells selected utilizing α/β CD3+/CD19+ cell depletion. All other treatment is standard of care.

DETAILED DESCRIPTION:
Patients wiith selected malignant or non-malignant conditions meeting eligibility criteria will be enrolled on this study. Patients will receive one of either full intensity, reduced intensity, or reduced toxicity conditioning appropriate based on disease, disease status, organ function and performance status and will undergo α/β T-cell and CD 19+ B cell depleted alloSCT.

Patients will be following for engraftment, chimerism, immune reconstitution, GVHD and QOL.

ELIGIBILITY:
Inclusion Criteria:

1. ALL:ALL high risk including one or more of the following: (t(9;22) or 11q23 chromosomal abnormality, primary induction failure (<15% blasts at time of registration), mixed phenotype acute leukemia (MPAL), persistent MRD (<0.01% by flow or persistent abnormal karyotype detected by cytogenetics) or hypodiploidy (44 chromosomes)) in first remission ' ALL in second remission and beyond;
2. AML: History of AML induction/reinduction Failure (<15% blasts at time of registration); AML in CR1 with poor cytogenetics (i.e. 12p, 5a, -7, FLT3 mutation/duplication, t(9;11) and others); AML with persistent minimal residual disease (MRD) in CR1(<0.01% on flow or persistent abnormal karyotype detected by cytogenetics); AML CR2 or beyond; AML in refractory relapse but ≤15% bone marrow leukemia blasts; Therapy-related AML
3. High Risk Myelodysplastic syndrome (MDS) 4 Lymphoma: Hodgkin (HL) or Non-Hodgkin (NHL): HL or NHL in induction failure; HL or NHL in PR1 or PR2 ; HL or NHL in CR2 or subsequent remission

5. Bone marrow failure syndromes: Kostmann syndrome refractory or intolerant to granulocyte colony-33stimulating factor; Diamond-Blackfan anemia refractory or intolerant to corticosteroids and/or cyclosporine'; amegakaryocytic thrombocytopenia 6. Sickle Cell Disease (Homozygous Hemoglobin S Disease, or Hemoglobin S β 0/+ thalassemia, or Hemoglobin SC Disease) 7. age 0-30 years 8. adequate organ function

Exclusion Criteria:

1. Females who are pregnant or breast-feeding are not eligible.
2. Patients with documented uncontrolled infection at the time of study entry are not eligible.
3. Karnofsky/Lansky (age appropriate) Performance Score <60
4. Demonstrated lack of compliance with medical care
5. Patients who have received allogeneic HSCT within 6 months, unless being done as a boost.
6. Patients with active <Grade 2 GVHD.

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events related to administration of α/β CD3+/CD19+ cell depleted stem cells | 1 year
  patients will be monitored for any adverse events related to administration of α/β CD3+/CD19+ cell depleted stem cells

SECONDARY OUTCOMES:
incidence of hematpoitic engraftment following Allogeneic stem cell transplantation (AlloSCT) utilizing α/β CD3+/CD19+ cell depletion | 1 year
  patients will have routine chimerism performed to monitoring engraftment of donor cells
incidence of GVHD following Allogeneic stem cell transplantation (AlloSCT) utilizing α/β CD3+/CD19+ cell depletion | 1 year
  patients will be monitored post transplant for signs of acute and chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, Study Chair — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No